CLINICAL TRIAL: NCT03606395
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Single Doses of NV-5138 in Healthy Volunteers and Subjects With Treatment-Resistant Depression
Brief Title: Safety, Tolerability, PK and Efficacy of Single Doses of NV-5138 in Healthy Volunteers and Subjects With Treatment-Resistant Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Navitor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAV-17A-001
Record Dates: First submitted 2018-07-10; First posted 2018-07-30 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — NV-5138

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, single dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single ascending dose_healthy subjects (Experimental): NV-5138:
  Single dose of 150, 300, 600, 1000, 1600 or 2400 mg single dose of placebo
  Interventions: Drug: NV-5138; Drug: Placebos
- Single dose in subjects with TRD (Experimental): NV-5138 oral solution single dose (dose to be determined from Part A) single dose of placebo
  Interventions: Drug: NV-5138; Drug: Placebos

INTERVENTIONS:
Drug: NV-5138 — single ascending dose
Drug: Placebos — Placebo liquid solution to mimic NV-5138

SUMMARY:
Randomized, two-part, placebo-controlled study of single ascending doses of NV-5138 in healthy volunteers, and a single dose of NV-5138 in subjects with Treatment-Resistant Depression (TRD)

DETAILED DESCRIPTION:
This is a randomized, two-part, double-blind, placebo-controlled study of single ascending dosage levels of NV-5138 in healthy volunteers and a single dose of NV-5138 in subjects with TRD. The study includes an up to 28-day screening period, an in-house period during which NV-5138 or placebo will be administered, and a 3- to 7-day follow-up period after discharge.

In Part A of the study (single-ascending-dose [SAD] portion in healthy volunteers), up to approximately 48 healthy volunteers will be randomly assigned to double-blind treatment. Eight (8) subjects will be randomized in each of six dosage-level cohorts (150, 300, 600, 1000, 1600, or 2400 mg NV-5138, or placebo, administered as an oral solution). Within each cohort, six subjects will be randomized to receive NV-5138 and two subjects will be randomized to receive placebo. Each subject will receive only one dose of either NV-5138 or placebo on Day 1. Within each cohort, initially one subject will receive NV-5138 and one subject will receive placebo. Provided no clinically significant safety issues are noted in the 24 hours after dosing the initial two subjects in the cohort, the six subjects remaining in the cohort may be dosed.

In Part B of the study (single-dose portion in subjects with TRD), up to approximately 40 subjects will be randomly assigned to double-blind treatment in one cohort. The dosage level for this cohort will be determined based on the safety, tolerability, and pharmacokinetic data from Part A of the study. However, in no case will the dose in Part B of the study exceed the highest dose administered in Part A of the study. Within this cohort, after potential eligibility has been confirmed by a site-independent review process, twenty (20) subjects will be randomized to receive NV-5138 and twenty (20) subjects will be randomized to receive placebo.

ELIGIBILITY:
Inclusion Criteria (Subjects in Part A or Part B):

1. Subjects must understand the nature of the study and must provide signed and dated written informed consent before the conduct of any study-related procedures.
2. Female subjects must be postmenopausal, surgically sterile, or agree to use one or more of the following forms of contraception from the time of signing the informed consent form through at least 30 days following the administration of test article: hormonal (i.e., oral, transdermal, implant, or injection); double barrier (i.e., condom, diaphragm with spermicide); intrauterine device (IUD); or vasectomized partner (6 months minimum). Postmenopausal women must have had ≥ 12 months of spontaneous amenorrhea with follicle-stimulating hormone [FSH] ≥ 30 mIU/mL. Surgically sterile women are defined as those who have had a hysterectomy, bilateral ovariectomy, or bilateral tubal ligation. All women must have a negative pregnancy test result before administration of test article.
3. Male subjects who are biologically capable of having children (i.e., non-vasectomized) must agree to use one or more of the above forms of birth control for either themselves or their partner(s), as appropriate, from the time of signing the informed consent form through at least 90 days following the administration of test article.
4. Subjects must be, in the opinion of the investigator, able to participate in all scheduled evaluations, likely to complete all required tests, and likely to be compliant.
5. Subjects must be fluent in English.

   Inclusion Criteria (Subjects in Part A Only):
6. Subjects must be age 18-55, inclusive.
7. Subjects must have a body mass index (BMI) between 19 and 30, inclusive.

   Inclusion Criteria (Subjects in Part B Only):
8. Subjects must be age 18-65, inclusive.
9. Subjects must have a BMI between 19 and 35, inclusive.
10. Subjects must have a diagnosis of major depressive disorder (MDD) without psychotic features, according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria, based on clinical assessment and confirmed by the Mini International Neuropsychiatric Interview (MINI).
11. Subjects must have had an inadequate response to at least one but no more than four antidepressants (stable, adequate dose, at least 6 weeks treatment) in the current episode of depression. The Massachusetts General Hospital-Antidepressant Treatment Response Questionnaire (MGH-ATRQ) will be used to assess antidepressant treatment response. Less than 50% improvement will be considered inadequate response.
12. Subjects must have a Montgomery-Åsburg Depression Rating Scale (MADRS) total score ≥ 21 at screen and at all evaluations between screen and dose administration (Day 1).
13. Subjects must have a Raskin Depression Rating Scale score ≥ 9 at screen and at all evaluations between screen and dose administration (Day 1).

Exclusion Criteria:

* Exclusion Criteria (Subjects in Part A or Part B):

Subjects must not have:

1. A positive pregnancy test result or be breastfeeding.
2. A clinically significant illness (including chronic, persistent, or acute infection), medical/surgical procedure, or trauma within 30 days prior to screen or between screen and dose administration (Day 1).
3. A history or presence of a clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, or neurologic abnormality.
4. A history or presence of any disease, condition, or surgery likely to affect drug absorption, distribution, metabolism, or excretion.
5. A clinically significant abnormality on physical examination, neurological examination, electrocardiogram (ECG), or laboratory evaluations at screen or between screen and dose administration (Day 1).
6. Alanine aminotransferase or aspartate aminotransferase levels greater than 1.5 times the upper limit of normal (ULN) at screen or between screen and dose administration (Day 1).
7. Creatinine clearance < 60 mL/min, according to the Cockcroft-Gault equation.
8. Leukocyte or neutrophil counts less than the lower limit of normal (LLN) at screen or between screen and dose administration (Day 1).
9. A clinically significant vital signs abnormality at screen or between screen and dose administration (Day 1). This includes, but is not limited to, the following, in the supine position (after 10 minutes supine controlled rest): (a) systolic blood pressure > 140 mmHg, (b) diastolic blood pressure > 90 mmHg, or (c) heart rate < 45 or > 85 beats per minute.
10. A corrected QT interval measurement corrected according to the Fridericia rule (QTcF) > 450 msec for men and > 470 msec for women during controlled rest at screen or between screen and dose administration (Day 1), or family history of long-QT syndrome.
11. Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG and any abnormalities in the 12-lead ECG that, in the judgement of the investigator, may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology or left ventricular hypertrophy.
12. PR (PQ) interval shortening < 120 msec (PR < 120 msec but > 110 msec is acceptable if there is no evidence of ventricular pre-excitation).
13. PR (PQ) interval prolongation (> 240 msec), intermittent second-degree (Wenckebach block while asleep or in deep rest is not exclusionary) or third-degree atrioventricular block.
14. Persistent or intermittent complete bundle branch block (BBB), or intraventricular conduction delay (IVCD) with QRS > 110 msec. Subjects with QRS > 110 msec but < 115 msec are acceptable if there is no evidence of ventricular hypertrophy or pre-excitation.
15. Significant (> 10%) weight loss or gain within 30 days prior to screen or between screen and dose administration (Day 1).
16. A history of seizure.
17. A history of clinically significant head trauma, including closed head injury with loss of consciousness.
18. A history of clinically significant symptomatic orthostatic hypotension (i.e., postural syncope).
19. A history of neuroleptic malignant syndrome.
20. A history of chronic urinary tract infections.
21. A history of cancer within 5 years prior to screen or between screen and randomization (with the exception of non-metastatic basal and/or squamous cell carcinoma of the skin), any history of renal cell carcinoma or breast cancer, or a family history of lymphangioleiomyomatosis in association with tuberous sclerosis complex (TSC-LAM).
22. Any illness or condition that, in the opinion of the investigator, (a) significantly increases the potential risk associated with the subject's participation in the study, (b) decreases the likelihood the subject will complete the study, and/or (c) may confound the results of the study.
23. A diagnosis of intellectual disability (intellectual developmental disorder) or mental retardation.
24. Used prescription or nonprescription medications for attention-deficit hyperactivity disorder (ADHD), narcolepsy, or cognitive enhancement (e.g., methylphenidate, atomoxetine, modafinil, ginkgo biloba, and huperzine A) within 1 month prior to screen or between screen and dose administration (Day 1).
25. Used any vitamin or herbal supplement within 2 weeks prior to dose administration (Day 1), unless approved by the investigator and medical monitor.
26. Consumed alcohol or used any over-the-counter medication (other than up to 3 g per day paracetamol/acetaminophen) within 7 days prior to screen or between screen and dose administration (Day 1).
27. Regularly consumed (e.g., more days than not) excessive quantities of xanthine-containing beverages (e.g., more than five cups of coffee or the equivalent per day) within 30 days prior to screen or between screen and dose administration (Day 1).
28. Donated blood or plasma within 6 weeks prior to screen or between screen and dose administration (Day 1).
29. Used any experimental medication, device, or biologic within 3 months or five half-lives (whichever is longer) prior to screen or between screen and dose administration (Day 1).
30. Currently employed by Navitor Pharmaceuticals, Inc. or by a clinical trial site participating in this study, or a first-degree relative of a Navitor Pharmaceuticals, Inc. employee or of an employee at a participating clinical trial site.
31. Any condition that, in the opinion of the investigator or medical monitor, makes the subject unsuitable for the study.
32. Strenuous physical activity within 1 week prior to dose administration (Day 1).
33. Unsatisfactory venous access.
34. Known or suspected hypersensitivity or idiosyncratic reaction to study drug or study drug excipients.

    Exclusion Criteria (Subjects in Part A Only):
35. A clinically significant abnormality on electroencephalogram (EEG) at screen (e.g., epileptiform activity).
36. Urine drug screen positive for a drug of abuse.
37. Used any prescription drug within 2 weeks prior to screen, or between screen and dose administration (Day 1).
38. Frequently used any tobacco-containing (e.g., cigar, cigarette or snuff) or nicotine-containing product (e.g., nicotine chewing gum, nicotine plasters, or other product used for smoking cessation) within 3 months prior to screen. Frequent use is defined as 3 or more days per week. Use of any tobacco- or nicotine-containing product is prohibited within 1 week of dose administration (Day 1).
39. Any history of psychiatric disorders, including substance use disorders, according to the DSM-5 criteria.
40. Acute suicidality as evidenced by answering "yes" for Question 4 ("Lifetime") or Question 5 ("Lifetime") on the Columbia-Suicide Severity Rating Scale (C-SSRS), indicating active suicidal ideation with any intent to act, at screen or between screen and dose administration (Day 1), or by answering "yes" for Question 3 ("In the Past Month") on the C-SSRS, indicating active suicidal ideation with any methods (not plan) without intent to act, at screen or between screen and dose administration (Day 1).
41. History of suicidal behavior such that a determination of "yes" is made on the Suicidal Behavior section of the C-SSRS for "Actual Attempt," "Interrupted Attempt," "Aborted Attempt," or "Preparatory Acts or Behavior."

    Exclusion Criteria (Subjects in Part B Only):
42. Urine drug screen positive for a drug of abuse, except cannabis. Prior use of cannabis is permitted provided the subject agrees to abstain from smoking or ingesting cannabis within 1 week of dose administration (Day 1) and during the study (including the follow-up period), and provided that, in the judgement of the investigator, the subject is likely to be compliant regarding this restriction.
43. Used any psychopharmacologic drug within 2 weeks prior to dose administration (Day 1), except for sleep medication, if used less than 4 days/week within 1 month prior to screen and between screen and dose administration (Day 1).
44. Any history of a psychotic disorder, MDD with psychosis, bipolar or related disorders, post-traumatic stress disorder, obsessive-compulsive disorder (if primary), intellectual disability (DSM-5 diagnostic code 319), borderline personality disorder, antisocial personality disorder, histrionic personality disorder, or narcissistic personality disorder, according to the DSM-5 criteria, or any other psychiatric or neurologic disorder or symptom that could pose undue risk to the subject or compromise the study.
45. Moderate or severe substance use disorder within 1 year prior to screen, according to the DSM-5 criteria.
46. Acute suicidality as evidenced by answering "yes" for Question 4 ("In the Past Year") or Question 5 ("In the Past Year") on the C-SSRS, indicating active suicidal ideation with any intent to act, at screen or between screen and dose administration (Day 1), or by answering "yes" for Question 3 ("In the Past Month") on the C-SSRS, indicating active suicidal ideation with any methods (not plan) without intent to act, at screen or between screen and dose administration (Day 1).
47. History of suicidal behavior such that a determination of "yes" is made on the Suicidal Behavior section of the C-SSRS ("In the Past Year") for "Actual Attempt," "Interrupted Attempt," "Aborted Attempt," or "Preparatory Acts or Behavior."
48. MADRS item 10 score of 5 at screen or between screen and dose administration (Day 1).
49. MADRS total score change ≥ 20% between screen and dose administration (Day 1).
50. Covi Anxiety scale score ≥ Raskin Depression Rating Scale score at screen or between screen and dose administration (Day 1).
51. History of clinically significant physical, sexual, or psychological abuse (age ≤ 7 years).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-06-09 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events as evidenced by CTCAE v.5.0 | Baseline through Day 9
  Number of subjects with treatment emergent adverse events

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of a single dose of NV-5138 | baseline to Day 4
  Maximum plasma concentration (Cmax)
Terminal elimination half-life (t1/2λz) of a single dose of NV-5138 | baseline to day 4
  Terminal elimination half-life (t1/2λz)
Area under the plasma concentration-time curve from zero to infinity (AUC) of a single dose of NV-5138 | baseline to day 4
  Area under the plasma concentration-time curve from zero to infinity (AUC)
Plasma clearance (CL) of a single dose of NV-5138 | baseline to day 4
  Plasma clearance (CL)
Mean residence time (MRT) of a single dose of NV-5138 | baseline to day 4
  Mean residence time (MRT)
change from baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score | baseline to Day 2
  The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition. The MADRS evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, inability to feel (interest level), pessimistic thoughts and suicidal thoughts.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Shelton, MD, Principal Investigator — University of Alabama at Birmingham
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Collaborative Neuroscience Network, Long Beach, California
  - Synergy San Diego, San Diego, California
  - MD Clinical, Hallandale, Florida
  - Innovative Clinical Research Inc, Hialeah, Florida
  - Research Centers of America, Hollywood, Florida
  - St. Louis Clinical Trials, St Louis, Missouri
  - Hassman Research Institute, Berlin, New Jersey
  - Midwest Clinical Research, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Targum SD, Sanacora G, Formella AE, Ceresoli-Borroni G, Owen R. A novel, experimental design to assess rapid antidepressant action: Results from a phase 1b randomized trial of NV-5138. J Psychiatr Res. 2026 Mar;194:211-220. doi: 10.1016/j.jpsychires.2026.01.006. Epub 2026 Jan 7. PMID 41512716